CLINICAL TRIAL: NCT03529734
Title: Evaluation of Neuro-Muscular Trunk Stabilization Functions and Development of Exercise Programs for Lower Back Pain Prevention
Brief Title: Changes in Trunk Stability Indicators Following Two Types of Exhausting Physical Activities
Acronym: TNC-FAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Primorska (Other)
Collaborators: S2P, Science to Practice, Ltd. (Other); Motus Melior (Unknown)
Responsible Party: Principal Investigator, Nejc Sarabon, Assoc. Prof. Dr. Sc., University of Primorska
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UP-FVZ-Fatigue&TrunkStability
Record Dates: First submitted 2018-02-12; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Spine Stiffness; Spine Stability
Keywords: Anticipatory postural adjustments; Trunk muscles reflex responses; Sitting balance; Kinesthesia
MeSH Terms: interventions — Running

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12 min running group (Experimental): This group will perform a 12 min high intensity running with the goal to cover maximal possible distance.
  Interventions: Other: 12 min running
- Local strengthening exercise group (Experimental): This group will perform local strengthening exercises (curl-ups, left side trunk flexion, trunk extension, right side trunk flexion). Each participant will have to perform three sets of each exercise with the maximal possible number of repetitions with a slow tempo (1s concentric phase and 2 s eccentric phase). Between sets, minimal rest (15 s) will be administered.
  Interventions: Other: Local strengthening exercises

INTERVENTIONS:
Other: 12 min running — This was already explained in the description of arm
  Arms: 12 min running group
Other: Local strengthening exercises — This was already explained in the description of arm
  Arms: Local strengthening exercise group

SUMMARY:
In this research project, effects of two sports specific types of fatiguing protocols on trunk muscles and specific trunk stability indicators will be studied. In general, sports activities involving gross motor activities activate higher percentage of muscle mass. In addition, such activities usually demand increased ventilation and more demanding inter-muscular activation. Such an example is running, with medium intensity until exhaustion or with the goal to cover the longest distance possible in a given time. On the contrary, sports practice often incorporates local strengthening exercises into a workout, especially for the trunk muscles. These, if performed correctly, cause localized muscle fatigue and can affect their function. Understanding the effects of these activities is of importance for coaches as well as for health care providers, as other types of training usually follow such activities that can more easily lead to trunk or spinal overload. We expect that localized muscle strengthening protocol until exhaustion will have more detrimental effects on trunk stability indicators as fatiguing with exhaustive running.

In these study 100 subjects will be studied, divided into two groups. First group will perform an exhaustive running protocol and the second group a localized trunk muscle strengthening protocol until exhaustion. The effect of intervention will be studied by observing the changes in trunk muscle reflex responses following sudden arm loading and changes in anticipated trunk muscle activation during a quick arm raising task. Activation latencies and electromyographic (EMG) amplitude, and center of foot pressure excursion will be used to quantify trunk stability. In addition, center of pressure movement during a sitting balance task will be studied as to gather information of local trunk stabilization functions. Finally, changes in joint position sense will be assessed in order to account for the possible changes in kinesthesia.

DETAILED DESCRIPTION:
It has been shown, that fatiguing a muscles in a kinetic chain leads to changes in activities of other non-fatigued muscles during postural tasks. This indicates that central changes take place to adapt the muscle responses according to the new state of the kinetic chain. However, these studies have mainly been focused on studying the effects of localized isometrically induced muscular fatigue that is less relevant to the sport community. In sports training, trunk muscle fatigue is often induced by performing dynamic strength training during a workout session, followed by other training interventions that pose high demands on trunk stability. On the other hand, more complex and gross motor tasks are used such as running, that also have the potential to influence trunk stability. Their effect on trunk stability comes from changes in muscle function as well as form increased ventilation. In both cases, trunk stability can be affected, leading to increased risk of injury. Especially the localized fatigue of the trunk muscles can have a direct effect on trunk stabilizing activities. One might speculate, that the intramuscular coordination can change as to compensate for the decreased ability of the trunk muscles to produce trunk and spinal stabilization impulses. After exhaustive running, especially trunk extensors might be affected, because of the increased trunk forward lean. In addition, trunk muscles are important contributors to increased ventilation in such tasks. As opposed to isolated fatiguing, running might have more complex effects on the trunk stabilization.

It is of most relevance for sports trainers and health care community dealing with athletes to be familiar with the effects of exhaustive running and localized trunk muscle fatigue on trunk and spinal stability in order to be better suited in preventing low back pain. This understanding will enable preparation of more suited training plans, periodization and individualization approaches.

This study will recruit volunteers form local university. Each participant will receive his own identification code that will be known only to the principal investigator. In order to account for the possible bias of the investigators, these will not be allowed to participate in assessing subject, which they are familiar with. Six investigators will participate, all trained in performing the measurement and fatiguing protocols.

All participants will be familiarized with the measurement tasks to overcome possible misunderstandings during the study and to ensure most fluent execution of the measurement protocol. The familiarization will account for as much time as needed for the participants to become proficient in each assessment task. Each participant will sigh an informed consent form that will be prepared in accordance with declaration of Helsinki.

Prior to starting the measurements, each subject will perform a worm-up. The measurement will follow in a predefined order, starting with the EMG electrode placement. First subjects will (ii) perform measurements of trunk muscles reflex responses during a sudden hand loading, followed by (iii) measurements of anticipatory postural adjustments during a quick arm rising test, (iv) body sway during a sitting balance tasks, (v) joint position test and (vi) measurements of maximal voluntary contraction for trunk extension and flexion in a neutral upright stance. Next, subjects will perform a fatiguing protocol. One group of subjects will perform a twelve-minute running test (Coopers test) with the goal to cower as much distance as possible. Subjects in the second group will perform dynamic strengthening exercises (curl-up, right lateral trunk flexion, trunk extension and left lateral trunk flexion), each session performed until exhaustion. All together subjects in a dynamic strengthening group will perform three sets with minimal rest in between. Immediately after finishing the fatiguing protocol, the above measurement protocol will be repeated in the same order.

The measurement data will be saved to a personal computers encoded with the subject's identification code. During data acquisition, processing, statistical analysis and data presentation only identification codes will be used. No individual data will be presented. All data will be gathered in a common data sheet for further statistical analysis.

Prior to performing the study, the sample size will be calculated based on the effect size of data gathered during a pilot study using 10 subjects. For main results, fallowing statistics will be calculated:

* Descriptive statistics.
* For parameters not normally distributed, appropriate corrections will be made.
* Intra-group differences prior to fatiguing protocol will be identified using the T-test for independent samples.
* For parameters, where no baseline differences between the two groups were observed, a Two-way repeated measures ANOVA model will be used to observe the possible changes after fatiguing protocols and possible interaction effects for the two groups. Observed differences will be additionally studied with post-hock tests.
* In cases where the baseline status between the two groups will be different, ANCOVA model will be used.
* Correlations between the parameters will be studied using Pearson correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age between 20 and 30 years

Exclusion Criteria:

* Chronic illness of the loco-motor system
* Acute injury of the loco-motor system in the last 1.5 years
* Neurological disease or injury
* Balance related pathology
* Vision pathology or untreated vision deficits

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Amplitude of EMG response to sudden arm raising. | Change from baseline to after intervention (12 minutes).
  EMG responses of the Erector spinae, Multifidus, Obliquus internus, Obliquus externus and Rectus abdominis will be studied.
Latency of EMG response to sudden arm raising. | Change from baseline to after intervention (12 minutes).
  EMG responses of the Erector spinae, Multifidus, Obliquus internus, Obliquus externus and Rectus abdominis will be studied.
Amplitude of EMG response to sudden arm loading. | Change from baseline to after intervention (12 minutes).
  EMG responses of the Erector spinae, Multifidus, Obliquus internus, Obliquus externus and Rectus abdominis will be studied.
Latency of EMG response to sudden arm loading. | Change from baseline to after intervention (12 minutes).
  EMG responses of the Erector spinae, Multifidus, Obliquus internus, Obliquus externus and Rectus abdominis will be studied.
Average Center of pressure velocity during sitting balance task. | Change from baseline to after intervention (12 minutes).
  Subjects will sit on an wobble board, that will be positioned on a force plate. The legs will be positioned on a specially designed rests mounted to the wobble board. Different parameters will be used to analyze the center of pressure movement (CoP), such as Average velocity of the CoP movement in both directions, Average amplitude and maximal amplitude in both directions and average frequency of CoP movement in both directions.
Average Center of pressure amplitude during sitting balance task. | Change from baseline to after intervention (12 minutes).
  Subjects will sit on an wobble board, that will be positioned on a force plate. The legs will be positioned on a specially designed rests mounted to the wobble board. Different parameters will be used to analyze the center of pressure movement (CoP), such as Average velocity of the CoP movement in both directions, Average amplitude and maximal amplitude in both directions and average frequency of CoP movement in both directions.
Average Center of Pressure frequency during sitting balance task. | Change from baseline to after intervention (12 minutes).
  Subjects will sit on an wobble board, that will be positioned on a force plate. The legs will be positioned on a specially designed rests mounted to the wobble board. Different parameters will be used to analyze the center of pressure movement (CoP), such as Average velocity of the CoP movement in both directions, Average amplitude and maximal amplitude in both directions and average frequency of CoP movement in both directions.
Trunk Reposition Error | Change from baseline to after intervention (12 minutes).
  Subjects will be standing upright with their eyes cowered. They will have to move into trunk flexion and hold a certain position determined by the investigator. In the next repetition the subject will have to repeat the same forward lean and hold the previously determined position. The parameter observed will be the difference between the angles.

SECONDARY OUTCOMES:
Maximal trunk extension voluntary torque | Change from baseline to after intervention (12 minutes).
  Subjects will be standing next to the custom designed dynamometer, measuring force in a neutral upright stance. During each repetition, an maximal force average over 1s interval will be calculated and used for further analysis.
Maximal trunk flexion voluntary torque | Change from baseline to after intervention (12 minutes).
  Subjects will be standing next to the custom designed dynamometer, measuring force in a neutral upright stance. During each repetition, an maximal force average over 1s interval will be calculated and used for further analysis.
Center of pressure velocity during sudden arm raising. | Change from baseline to after intervention (12 minutes).
  During quick hand rising task, subjects will be standing on a force plate. Amplitude of the Center of pressure movement will be analyzed 150 ms before and 150 ms after EMG onset.
Center of pressure amplitude during sudden arm raising. | Change from baseline to after intervention (12 minutes).
  During quick hand rising task, subjects will be standing on a force plate. Amplitude of the Center of pressure movement will be analyzed 150 ms before and 150 ms after EMG onset.
Center of pressure velocity during sudden arm loading. | Change from baseline to after intervention (12 minutes).
  During sudden hand loading task subjects will be standing on a force plate. Center of pressure movement will be analyzed 250 ms after loading the hands.
Center of pressure amplitude during sudden arm loading. | Change from baseline to after intervention (12 minutes).
  During sudden hand loading task subjects will be standing on a force plate. Center of pressure movement will be analyzed 250 ms after loading the hands.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No